CLINICAL TRIAL: NCT01701817
Title: Outcomes Registry for Better Informed Treatment of Atrial Fibrillation II (Orbit-AF II)
Acronym: ORBIT-AF II
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Duke Clinical Research Institute (Other); Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100871; RIVAROXAFL4002 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Irregular heart beat
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Atrial Fibrillation (AF): (1) patients with new onset/first detected Atrial Fibrillation (AF) diagnosed within the 6 months preceding the baseline visit; or (2) patients with AF who had initiation or transition to a FXa (Factor Xa) inhibitor or a direct thrombin inhibitor within the preceding 3 months.
  Interventions: Other: Patients with Atrial Fibrillation

INTERVENTIONS:
Other: Patients with Atrial Fibrillation — Treatment patterns of AF according to patient demographics, clinical factors, risk stratification, and geographic regions.

SUMMARY:
The Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF II) is a multicenter, prospective outpatient disease registry to evaluate the utilization of target-specific antithrombotic agents, such as FXa (factor Xa) inhibitors and direct thrombin inhibitors, and associated outcomes. Importantly, the ORBIT AF II registry will permit the collection and analysis of post-approval observational data needed for evaluating the outcomes associated with these new agents when used in broader patient populations outside of clinical studies. The ORBIT-AF II registry will focus on patients with newly diagnosed atrial fibrillation (AF) as well as those who have been recently started on a target-specific oral anticoagulant agent. Taken together, the ORBIT-AF I and ORBIT-AF II registries will offer a broad and contemporary view of AF therapy.

DETAILED DESCRIPTION:
The registry will be used to evaluate, describe, and document the safety of target-specific anticoagulant agents (and other antithrombotic agents) in patients with Atrial Fibrillation (AF), the clinical outcomes associated with their use, the treatment patterns and clinical course of patients with AF, including those who undergo cardiac procedures of interest (ablation, cardioversion, catheterization and surgery, for examples), and characteristics of patients with new onset/first-detected AF. Additionally, the registry will be used to summarize patterns of switching or discontinuation of antithrombotic agents in the United States. The registry will be a nationwide collaboration of health care providers (eg, cardiologists, internists, primary care physicians, electrophysiologists, quality improvement personnel, office/practice managers, research coordinators, and pharmacists). Target enrollment will be approximately 15,000 patients. It is anticipated that enrollment will complete in approximately 3.5 years. Consecutive patients who meet the eligibility criteria will be approached and educated about the registry. Patients who express interest will provide informed consent. Patients enrolled in the registry will be followed for up to 2 years. New patients enrolled in the registry will be followed for up to 1 year. Patient follow-up by their AF care provider will continue as scheduled according to local clinical practice. Data collection will occur at 6 month intervals for approximately 1 year from the time of enrollment of the patient (baseline, 6, and 12 months). Data capture will include demographics, medical history, cardiovascular history, vital signs, echocardiographic and laboratory data, AF status and type (paroxysmal, persistent, long-standing persistent/permanent), pharmacotherapy, contraindications to oral anticoagulant therapy, and provider specialty. Clinical outcomes and safety data capture will include major adverse cardiac events (MACEs).

ELIGIBILITY:
Inclusion Criteria: - Adult patients with incident (initial diagnosis) AF (Atrial Fibrillation) with electrocardiographic documentation or patients with prevalent (existing diagnosis) AF who had initiation or transition to a FXa (Factor Xa) inhibitor or a direct thrombin inhibitor within the preceding 3 months - anticipated ability to adhere to local regularly scheduled follow-up visits

-

Exclusion Criteria:

* Atrial flutter only - Anticipated life expectancy less than 6 months - short lasting AF secondary to a reversible condition (e.g. hyperthyroidism, pulmonary embolism, post-cardiothoracic surgery) - Participation in a randomized trial of anticoagulation for AF at the time of enrollment - Was enrolled in the ORBIT-I Registry

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolling physicians will include cardiologists, internists, and electrophysiologists from both academic and private practice who preferably have experience in registry participation.
Sampling Method: Non-Probability Sample
Enrollment: 13769 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Number of major bleeding events | 2 years
  Major bleeding will be defined according to International Society of Thrombosis and Hemostasis (ISTH) criteria.

SECONDARY OUTCOMES:
Number of major adverse cardiac events | 2 years
  Major cardiac events are defined as stroke or non-central nervous system (non-CNS) systemic embolism, myocardial infarction, and cardiovascular death.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (219):
- United States (217):
  - Cullman, Alabama
  - Dothan, Alabama
  - Fairhope, Alabama
  - Mobile, Alabama
  - Tuscaloosa, Alabama
  - Avondale, Arizona
  - Glendale, Arizona
  - Goodyear, Arizona
  - Scottsdale, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Alhambra, California
  - Anaheim, California
  - Bakersfield, California
  - Banning, California
  - Beverly Hills, California
  - Carlsbad, California
  - Concord, California
  - East Palo Alto, California
  - Fresno, California
  - Huntington Beach, California
  - Laguna Hills, California
  - Larkspur, California
  - Long Beach, California
  - Los Alamitos, California
  - Los Angeles, California
  - Manhattan Beach, California
  - Mission Hills, California
  - Newport Beach, California
  - Northridge, California
  - Pasadena, California
  - Pismo Beach, California
  - Pomona, California
  - Poway, California
  - Rancho Mirage, California
  - San Pedro, California
  - Santa Rosa, California
  - Torrance, California
  - Ventura, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Bridgeport, Connecticut
  - Guilford, Connecticut
  - Laurel, Delaware
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Bay Pines, Florida
  - Clearwater, Florida
  - Coral Springs, Florida
  - Eustis, Florida
  - Jupiter, Florida
  - Lakeland, Florida
  - Miami, Florida
  - Miramar, Florida
  - Palm Harbor, Florida
  - Pensacola, Florida
  - Port Charlotte, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Alpharetta, Georgia
  - Athens, Georgia
  - Atlanta, Georgia
  - Cumming, Georgia
  - Gainesville, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Rome, Georgia
  - Smyrna, Georgia
  - Idaho Falls, Idaho
  - Pocatello, Idaho
  - Aurora, Illinois
  - Hines, Illinois
  - Melrose Park, Illinois
  - New Lenox, Illinois
  - North Chicago, Illinois
  - Peoria, Illinois
  - Rock Island, Illinois
  - Anderson, Indiana
  - Bloomington, Indiana
  - Hammond, Indiana
  - Indianapolis, Indiana
  - La Porte, Indiana
  - Munster, Indiana
  - South Bend, Indiana
  - Davenport, Iowa
  - Waterloo, Iowa
  - Overland Park, Kansas
  - Elizabethtown, Kentucky
  - Louisville, Kentucky
  - Mount Sterling, Kentucky
  - Alexandria, Louisiana
  - Bossier City, Louisiana
  - Natchitoches, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Rockport, Maine
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Randallstown, Maryland
  - Salisbury, Maryland
  - Fall River, Massachusetts
  - Alpena, Michigan
  - Bay City, Michigan
  - Flint, Michigan
  - Grand Blanc, Michigan
  - Lansing, Michigan
  - Lapeer, Michigan
  - Mount Clemens, Michigan
  - Rochester Hills, Michigan
  - Saint Joseph, Michigan
  - Traverse City, Michigan
  - Troy, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Bridgeton, Missouri
  - Kansas City, Missouri
  - Fremont, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Nashua, New Hampshire
  - Bridgewater, New Jersey
  - East Brunswick, New Jersey
  - Flemington, New Jersey
  - Linden, New Jersey
  - Manalapan, New Jersey
  - Moorestown, New Jersey
  - Mountain Lakes, New Jersey
  - Somerset, New Jersey
  - Toms River, New Jersey
  - Voorhees Township, New Jersey
  - Wayne, New Jersey
  - Albany, New York
  - Flushing, New York
  - Huntington, New York
  - Jackson Heights, New York
  - Jamaica, New York
  - Jamestown, New York
  - Lake Success, New York
  - Mineola, New York
  - Mount Kisco, New York
  - New York, New York
  - North Massapequa, New York
  - Utica, New York
  - Burlington, North Carolina
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Elizabeth City, North Carolina
  - Greensboro, North Carolina
  - Pinehurst, North Carolina
  - Sanford, North Carolina
  - Spartanburg, North Carolina
  - Canton, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mansfield, Ohio
  - Miamisburg, Ohio
  - Toledo, Ohio
  - Worthington, Ohio
  - Youngstown, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Abington, Pennsylvania
  - Chambersburg, Pennsylvania
  - Doylestown, Pennsylvania
  - Ephrata, Pennsylvania
  - Langhorne, Pennsylvania
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sayre, Pennsylvania
  - West Reading, Pennsylvania
  - Wynnewood, Pennsylvania
  - Yardley, Pennsylvania
  - Providence, Rhode Island
  - Warwick, Rhode Island
  - Woonsocket, Rhode Island
  - Charleston, South Carolina
  - Easley, South Carolina
  - Lancaster, South Carolina
  - Bristol, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Oak Ridge, Tennessee
  - Austin, Texas
  - Beaumont, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Katy, Texas
  - McKinney, Texas
  - Odessa, Texas
  - Palestine, Texas
  - Plano, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Tyler, Texas
  - Annandale, Virginia
  - Lynchburg, Virginia
  - Mechanicsville, Virginia
  - Midlothian, Virginia
  - Newport News, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - Walla Walla, Washington
  - Charleston, West Virginia
  - La Crosse, Wisconsin
  - Milwaukee, Wisconsin
  - Waukesha, Wisconsin
  - Wausau, Wisconsin
- Río Grande, Puerto Rico
- Charlotte Amalie, Virgin Islands

REFERENCES:
- [Derived] Fox KAA, Virdone S, Pieper KS, Bassand JP, Camm AJ, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Kayani G, Oto A, Misselwitz F, Piccini JP, Dalgaard F, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. GARFIELD-AF risk score for mortality, stroke, and bleeding within 2 years in patients with atrial fibrillation. Eur Heart J Qual Care Clin Outcomes. 2022 Mar 2;8(2):214-227. doi: 10.1093/ehjqcco/qcab028. PMID 33892489
- [Derived] Jackson LR 2nd, Kim S, Blanco R, Thomas L, Ansell J, Fonarow GC, Gersh BJ, Go AS, Kowey PR, Mahaffey KW, Hylek EM, Peterson ED, Piccini JP; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation II. Discontinuation rates of warfarin versus direct acting oral anticoagulants in US clinical practice: Results from Outcomes Registry for Better Informed Treatment of Atrial Fibrillation II (ORBIT-AF II). Am Heart J. 2020 Aug;226:85-93. doi: 10.1016/j.ahj.2020.04.016. Epub 2020 Apr 28. PMID 32526533
- [Derived] Jackson LR 2nd, Kim S, Fonarow GC, Freeman JV, Gersh BJ, Go AS, Hylek EM, Kowey PR, Mahaffey KW, Singer D, Thomas L, Blanco R, Peterson ED, Piccini JP Sr; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation Patients and Investigators. Stroke Risk and Treatment in Patients with Atrial Fibrillation and Low CHA2DS2-VASc Scores: Findings From the ORBIT-AF I and II Registries. J Am Heart Assoc. 2018 Aug 21;7(16):e008764. doi: 10.1161/JAHA.118.008764. PMID 30369317
- [Derived] Inohara T, Kim S, Pieper K, Blanco RG, Allen LA, Fonarow GC, Gersh BJ, Ezekowitz MD, Kowey PR, Reiffel JA, Naccarelli GV, Chan PS, Mahaffey KW, Singer DE, Freeman JV, Steinberg BA, Peterson ED, Piccini JP; ORBIT AF Patients and Investigators. B-type natriuretic peptide, disease progression and clinical outcomes in atrial fibrillation. Heart. 2019 Mar;105(5):370-377. doi: 10.1136/heartjnl-2018-313642. Epub 2018 Sep 18. PMID 30228248
- [Derived] Steinberg BA, Shrader P, Pieper K, Thomas L, Allen LA, Ansell J, Chan PS, Ezekowitz MD, Fonarow GC, Freeman JV, Gersh BJ, Kowey PR, Mahaffey KW, Naccarelli GV, Reiffel JA, Singer DE, Peterson ED, Piccini JP; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) II Investigators. Frequency and Outcomes of Reduced Dose Non-Vitamin K Antagonist Anticoagulants: Results From ORBIT-AF II (The Outcomes Registry for Better Informed Treatment of Atrial Fibrillation II). J Am Heart Assoc. 2018 Feb 16;7(4):e007633. doi: 10.1161/JAHA.117.007633. PMID 29453305
- [Derived] Kaufman BG, Kim S, Pieper K, Allen LA, Gersh BJ, Naccarelli GV, Ezekowitz MD, Fonarow GC, Mahaffey KW, Singer DE, Chan PS, Freeman JV, Ansell J, Kowey PR, Rieffel JA, Piccini J, Peterson E, O'Brien EC. Disease understanding in patients newly diagnosed with atrial fibrillation. Heart. 2018 Mar;104(6):494-501. doi: 10.1136/heartjnl-2017-311800. Epub 2017 Aug 8. PMID 28790169
- [Derived] Steinberg BA, Shrader P, Thomas L, Ansell J, Fonarow GC, Gersh BJ, Hylek E, Kowey PR, Mahaffey KW, O'Brien EC, Singer DE, Peterson ED, Piccini JP; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Investigators and Patients. Factors associated with non-vitamin K antagonist oral anticoagulants for stroke prevention in patients with new-onset atrial fibrillation: Results from the Outcomes Registry for Better Informed Treatment of Atrial Fibrillation II (ORBIT-AF II). Am Heart J. 2017 Jul;189:40-47. doi: 10.1016/j.ahj.2017.03.024. Epub 2017 Apr 4. PMID 28625380
- [Derived] Steinberg BA, Simon DN, Thomas L, Ansell J, Fonarow GC, Gersh BJ, Kowey PR, Mahaffey KW, Peterson ED, Piccini JP; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Investigators and Patients. Management of Major Bleeding in Patients With Atrial Fibrillation Treated With Non-Vitamin K Antagonist Oral Anticoagulants Compared With Warfarin in Clinical Practice (from Phase II of the Outcomes Registry for Better Informed Treatment of Atrial Fibrillation [ORBIT-AF II]). Am J Cardiol. 2017 May 15;119(10):1590-1595. doi: 10.1016/j.amjcard.2017.02.015. Epub 2017 Mar 28. PMID 28363354
- [Derived] Steinberg BA, Shrader P, Thomas L, Ansell J, Fonarow GC, Gersh BJ, Kowey PR, Mahaffey KW, Naccarelli G, Reiffel J, Singer DE, Peterson ED, Piccini JP; ORBIT-AF Investigators and Patients. Off-Label Dosing of Non-Vitamin K Antagonist Oral Anticoagulants and Adverse Outcomes: The ORBIT-AF II Registry. J Am Coll Cardiol. 2016 Dec 20;68(24):2597-2604. doi: 10.1016/j.jacc.2016.09.966. PMID 27978942
- [Derived] Steinberg BA, Blanco RG, Ollis D, Kim S, Holmes DN, Kowey PR, Fonarow GC, Ansell J, Gersh B, Go AS, Hylek E, Mahaffey KW, Thomas L, Chang P, Peterson ED, Piccini JP; ORBIT-AF Steering Committee Investigators. Outcomes Registry for Better Informed Treatment of Atrial Fibrillation II: rationale and design of the ORBIT-AF II registry. Am Heart J. 2014 Aug;168(2):160-7. doi: 10.1016/j.ahj.2014.04.005. Epub 2014 Apr 18. PMID 25066554